CLINICAL TRIAL: NCT03693508
Title: Phase IV, Open, Multicentre, Single-arm Study to Evaluate the Efficacy and Safety of Elvitegravir / Cobicistat / Emtricitabine / Tenofovir Alafenamide as a First-line Treatment in Naïve Patients With HIV-1 Infection With Severe Immunosuppression.
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Elvitegravir / Cobicistat / Emtricitabine / Tenofovir Alafenamide as a First-line Treatment in Naïve Patients With HIV-1 Infection With Severe Immunosuppression
Acronym: GENIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 9216
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections; Severe Immunosuppression
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Single arm, phase 4 study. The naive patients will be treated with elvitegravir / cobicistat / emtricitabine / tenofovir alafenamide as a first-line treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Naive HIV patients with severe immunosuppression.
  Interventions: Drug: Genvoya®

INTERVENTIONS:
Drug: Genvoya® — Patents treated with elvitegravir (EVG) 150mg / cobicistat (COBI) 150mg / emtricitabine (FTC) 200mg / tenofovir (TAF) 10mg once a day as the first line treatment.
  Other Names: TAF/FTC/EVG-cb

SUMMARY:
Phase IV, open, multicentre and single-arm study. 50 HIV infection naive patients with severe immunosuppression will be recruited to evaluate the efficacy and safety of elvitegravir / cobicistat / emtricitabine / tenofovir alafenamide as a first-line treatment.

DETAILED DESCRIPTION:
The patients included in the study will be treated during 48 weeks and will have to perform the selection/basal visit, week 4 visit, week 8 visit, week 12 visit, week 24 visit, week 48 visit and follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give their written consent to participate in the study after having received information about the design, the purposes of the study, the possible risks that may arise from it and the possibility of withdrawing from it at any time. moment
* Adult patients (age ≥18 years) of both sexes
* Patients with HIV-1 infection with severe immunosuppression, defined by a concentration of CD4 + lymphocytes <200 cells / μL
* Patients who are allowed to perform a genotypic resistance test to inhibitors of intregrase, emtricitabine or tenofovir
* Creatinine clearance ≥ 30 ml / min before the start of treatment
* Alanine transaminase (ALT) / Aspartate transaminase (AST) levels not higher than five times normal levels, total bilirubin with normal values, neutrophils> 1000 cells / μL,> 50000 platelets / μL,> Hb level of 85 g / L and serum amylase levels <1 , 5 times higher normal limit before the start of treatment

Exclusion Criteria:

* Patient who undergoes a concomitant treatment not allowed. Patient with documented intolerance or hypersensitivity to the study medication, or who is contraindicated to use it, attending a technical file
* Patient receiving therapies with interferon, interleukin 2, cytotoxic chemotherapy or immunosuppressants at the baseline visit.
* Patients with neoplasms, an exception of skin cancer and anus cancer in situ (stage 0)
* Patient with any medical or psychological, sociological or geographical alteration, toxic habit (drugs, alcohol) that, a criterion of the researcher, may interfere in the fulfillment of the study by the patient. These conditions will be discussed with the patient before their inclusion in the trial
* Patients with any medical or psychological alteration that, a criterion of the investigator, an involuntary factor of the patient's ability to understand and complement the questionnaires and scales used in the study
* Patient in a treatment with any type of drug / product under investigation or who is participating in a clinical trial that uses a product under investigation, with the exception of studies in which the study treatment was completed more than 12 weeks ago
* Pregnant women, in breastfeeding period or with a positive pregnancy test in the selection period; women of childbearing age and sexually active who are not willing to use an adequate contraceptive method during the study and up to 3 months after the administration of the last dose of study treatment. Some women in adulthood have undergone permanent infertility procedures or amenorrheic procedures for less than 12 months
* Patients with severe hepatic impairment (Child-Pugh Class C).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with undetectable plasma viral load | Week 48
  study the effectiveness of the combination of TAF/FTC/EVG-cb

SECONDARY OUTCOMES:
Proportion of patients with virological failure | From basal until week 48
  Proportion of patients with Plasma viral load of HIV-1 RNA ≥50 copies / mL in the last measurement while the patient receives the treatment in the window period, patients who interrupt the treatment prematurely due to lack / loss of efficacy in which the last viral load was ≥50 copies / mL or in which the antiretroviral treatment was modified before 48 weeks.
Proportion of patients with virological failure | From basal visit until week 48
  Proportion of patients who interrupt the treatment prematurely due to absence or loss of efficacy
Proportion of patients with virological failure | From basal visit until week 48
  Proportion of patients who interrupt the treatment prematurely by others reasons (other than an adverse event, death or loss of effectiveness) and whose last viral load at the time of abandonment was ≥50 copies / mL.
Time to virological suppression | From basal until week 48
  viral load <50 copies / mL
Proportion of patients with virological failure while receiving antiretroviral treatment (ART), having previously been suppressed . | From basal until week 48
  virological failure defined by protocol as viral load> 1000 copies / mL at week 24 or 2 consecutive viral loads> 50 copies / mL (at least 2 weeks apart)
Time to virological failure | From basal until week 48
  Viral load ≥50 copias/mL
Incidence of genotypic resistance in patients with virological failure | From basal until week 48
Changes in viral load | Weeks 4, 8, 12, 24, 36 and 48
  plasma concentration of HIV RNA
Change in the CD4+ lymphocyte count | Week 48
Proportion of patients who have a CD4+ lymphocyte count > 200 cells / μL | Week 48
Mean time to reach a CD4 + lymphocyte count> 200 cells / μL | From basal until week 48

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Costa del Sol, Marbella, Malaga
  - H. Ramón y Cajal, Madrid
  - H. Clínico San Carlos, Madrid
  - H. Doce de Octubre, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No